CLINICAL TRIAL: NCT01340378
Title: A Pilot Study of Thrombin Generation Changes in Neonates Undergoing Placement of a Blalock-Taussig Shunt
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Children's healthcare of Atlanta: Cardiac Research Donor Funds (Unknown)
Responsible Party: Principal Investigator, Nina Guzzetta, M.D., Associate professor of Anesthesiology, Emory University
Other Study IDs: IRB00034496
Record Dates: First submitted 2011-04-12; First posted 2011-04-22 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Aortic Coarctation
Keywords: neonatal surgery; Blalock-Taussig shunt
MeSH Terms: conditions — Aortic Coarctation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples only
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary goal of this investigation is to describe perioperative thrombin generation in neonates undergoing placement of a Blalock-Taussig (BT) shunt to better understand the coagulation changes that precipitate postoperative shunt occlusion.

DETAILED DESCRIPTION:
To accomplish our goal, the investigators will measure preoperative levels of one major procoagulant (prothrombin) and one major anticoagulant (Antithrombin). The investigators will also measure preoperative and postoperative thrombelastograms (TEG) and preoperative and postoperative thrombin generation curves (TGC).

ELIGIBILITY:
Inclusion Criteria:

1. Full-term neonates (37-42 weeks gestational age)
2. Apgar score of 7 or more at 5 minutes after delivery
3. Surgical placement of BT shunt or repair of an aortic coarctation
4. Parent or legal guardian willing to participate, and able to understand and sign the provided informed consent

Exclusion Criteria:

1. Preterm neonates (less than 37 weeks gestation)
2. Apgar score of less than 7 at 5 minutes after birth
3. Emergent procedure
4. Surgical procedure other than placement of BT shunt or repair of aortic coarctation
5. Neonates with a known coagulation defect or coagulopathy
6. Mother with a known coagulation defect or coagulopathy
7. Parent or legal guardian unwilling to participate or unable to understand and sign the provided informed consent

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 1. Full-term neonates (37-42 weeks gestational age)
  2. Apgar score of 7 or more at 5 minutes after delivery
  3. Surgical placement of BT shunt or repair of an aortic coarctation
  4. Parent or legal guardian willing to participate, and able to understand and sign the provided informed consent
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Thrombin generation - peak amount | 2 years
  The thrombin generating capacity of plasma is measured using a fluorogenic substrate. Coagulation is initiated by contact activation and thrombin generation is monitored by a microplate fluorometer set that displays the progression of the fluorescence reaction. The peak amount of thrombin generated is expressed by absorbancy (nM).

SECONDARY OUTCOMES:
Thrombin Generation Curve validation in neonates | 2 years
  The peak amount of thrombin generated as determined by the thrombin generation curve will be compared to the peak amount of thrombin generated as determined by the thromboelastogram. Both measure thrombin generation by absorbancy (nM).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States